CLINICAL TRIAL: NCT06751082
Title: Sotatercept Pulmonary Hypertension Observational Registry
Brief Title: Real World Observational Study of Sotatercept for Pulmonary Hypertension
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert P. Frantz, Principal Investigator, Mayo Clinic
Other Study IDs: 24-011370
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study seeks to describe the real world initial experience with sotatercept in the treatment of pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or greater who are being treated with sotatercept in the Mayo Pulmonary hypertension clinic.

Exclusion Criteria:

* Adults lacking capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for whom sotatercept is being or has been prescribed will be identified through the Mayo Pulmonary Hypertension Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
EmPHasis10 Questionnaire | Baseline, Year 1, Year 2, Year 3, Year 4, Year 5, Year 6, Year 7, Year 8, Year 9, Year 10
  The EmPHasis10 Questionnaire consists of 10 questions to assess quality of life. The scores can range from 0-50, a higher score indicates a worse quality of life.
Number of pulmonary hypertension vasodilator medications taken by a subject | Baseline, Year 10
  Pulmonary hypertension vasodilator medications are used to decrease pressure in the pulmonary arteries.
Number of patients to have a change in dose of prostanoid medications | Baseline, Year 10
  A change in dose of prostanoid medications will be determined by a change from baseline dosage.
Number of patient hospitalizations | Baseline, Year 10
  Number of patient hospitalizations will be determined by the number of patients admitted into the hospital.
Number of patients to cease therapy sessions | Baseline, Year 10
  Cease of therapy session will be determined by a patient's termination of all therapy sessions
Number of patients to discontinue prostanoid therapy | Baseline, Year 10
  Number of patients to discontinue prostanoid therapy will be determined by a patients termination of all prostanoid therapy
Number of patients with bleeding complications | Baseline, Year 10
  Bleeding complications include nosebleeds not requiring ER visit or transfusion, epistaxis or GI hemorrhage requiring ED visit/hospitalization.
Number of patients to develop Skin telangiectasias | Baseline, Year 10
  Development of skin telangiectasias includes new development, worsening, or distribution
Change in 6 min walk distance | Baseline, Year 10
  6 minute walk distance will be measured in meters (m).
Number of patients to have a change in hemodynamics | Baseline, Year 10
  Change in hemodynamics include the change in Blood Flow, Blood Pressure, Cardiac Output, Vascular Resistance, Perfusion
Change in Right Ventricular Systolic Pressure (RVSP) | Baseline, Year 10
  Right Ventricular Systolic Pressure is the pressure in the right ventricle during contraction. RVSP will be measured in mmHg.
Right Ventricular Strain | Baseline, Year 10
  Right Ventricular Strain refers to strain on the right ventricle during contraction. Right Ventricular Strain will be determined by echocardiogram and measured as a percentage.
Change in Right Ventricle (RV) function | Baseline, Year 10
  Change in RV function will be determined by echocardiogram and measured as a percentage.
Change in capacitance | Baseline, Year 10
  Capacitance is the ability for blood vessels to store and release blood. capacitance will be determined by echocardiogram.
Change in tricuspid regurgitation | Baseline, Year 10
  Tricuspid regurgitation is the regurgitation of blood into the right atrium during contraction of the heart.
Change in Stroke Volume (SV) | Baseline, Year 10
  Stroke Volume is calculated by End-Diastolic Volume (EDV)-End-Systolic Volume (ESV) and measured in mL
Change in Pulse Pressure (PP) | Baseline, Year 10
  Pulse Pressure is calculated by PP=systolic blood pressure (SBP) - diastolic blood pressure (DBP) and measured in mmHg
Change in functional class | Baseline, Year 10
  Functional class refers to the severity of patients heart condition. A change in class would refer to the increase or decrease in severity of the condition.
Number of patients to survive without receiving a transplant | Baseline, Year 10
  A transplant is defined as receiving an organ or tissue from a donor.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Frantz, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No